CLINICAL TRIAL: NCT01123148
Title: A P300 Brain Computer Interface to Operate Power Wheelchair Tilt
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Jane Huggins, PhD, Research Assistant Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: M0001; R21HD054913 (NIH)
Record Dates: First submitted 2010-05-04; First posted 2010-05-14 (Estimated); Results first posted 2016-08-01 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-06

CONDITIONS: Healthy; Amyotrophic Lateral Sclerosis
Keywords: Brain computer interface; wheelchair control
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tilt testing (Other)
  Interventions: Device: Using a BCI to control wheelchair tilt

INTERVENTIONS:
Device: Using a BCI to control wheelchair tilt — Subjects will wear an EEG cap for 1-4 hours (1-2 hours typical) during each session and use a P300 based BCI to type words and control wheelchair tilt. Subjects will be asked to participate in 3 sessions.

SUMMARY:
The investigators want to develop a brain-computer interface (BCI) that will eventually allow people who are completely paralyzed to independently control the tilt feature on their power wheelchairs. This study will allow healthy volunteers to test the feasibility and accuracy of controlling a BCI using only their brain signals while seated in a tilting wheelchair.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older.
* Able to read text on a computer screen
* Able to understand and remember instructions concerning participation.

Exclusion Criteria:

* Unable give informed consent.
* Unable to understand and follow instructions.
* Have abnormal tone or uncontrolled movements in the head-and-neck that would interfere with EEG recordings.
* Known to have photosensitive epilepsy.
* Open head lesions or sores.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-01; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane Huggins, PhD, Principal Investigator — University of Michigan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 16 people consented, 2 were pilot subjects, not intended for inclusion in the final analysis. They helped to test the protocol and set-up for the planned data collection session to make sure that the instructions for future subjects were clear and that all equipment was working correctly.
Period: Overall Study
Arm/Group | Tilt Testing
Started | 14
BCI Calibration >50% Accuracy | 13
Completed | 12
Not Completed | 2
Not completed — Coughing caused unacceptable EEG quality | 1
Not completed — Didn't meet milestone criteria | 1

BASELINE CHARACTERISTICS:
Arm/Group | Tilt Testing
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 40.5 [19 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: The Accuracy of BCI Typing While Tilting in a Power Wheelchair and While Sitting Still in a Power Wheelchair.
Description: Subjects will participate in 3 sessions. During each session each subject will copy a "word" in each of 3 conditions (no-movement, self-movement, continuous movement) by typing using only brainwaves. For the no-movement condition, the wheelchair seat remains in a fixed position. For the self-movement condition, the angle of the wheelchair seat changes in response to some of the selections made with the brain-computer interface. For the continuous movement condition, the angle of the wheelchair seat moves continuously. Changes in the wheelchair's position may affect spelling accuracy. The accuracy of the subject's copy spelling of the designated word will be measured for each condition in each session. The order of the conditions is balanced across the three days. The accuracy for each subject in each condition is presented as the average of the accuracies for that condition across the three days.
Time Frame: 3 1-2 hour sessions over 2-4 weeks
Measure: Mean (Standard Deviation); unit: % Accuracy of selections
Arm/Group | Tilt Testing
Number analyzed (Participants) | 12
% Accuracy of selections
  No Movement | 91.04 (6.93)
  BCI Controlled Movement | 91.18 (6.36)
  Continuous Movement | 88.38 (11.69)

ADVERSE EVENTS:
Arm/Group | Tilt Testing
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

LIMITATIONS AND CAVEATS:
This study only includes data from able-bodied individuals.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No